CLINICAL TRIAL: NCT01563523
Title: A Multi-centre, Randomised, Double-blind, Parallel Group, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Activated Recombinant Factor VII (rFVIIa/NovoSeven®/ Niastase®) in the Treatment of Bleeding in Severely Injured Trauma Subjects
Brief Title: Efficacy and Safety of Activated Recombinant Human Factor VII in Severely Injured Trauma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7TRAUMA-2159
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activated recombinant human factor VII (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — Standard therapy in conjunction with three single doses of rFVIIa administered over a 3 hour period. Administered once the subject has received 8 units of PRBC
  Arms: Activated recombinant human factor VII
Drug: placebo — Standard therapy in conjunction with three single doses of placebo administered over a 3 hour period. Administered once the subject has received 8 units of PRBC
  Arms: Placebo

SUMMARY:
This trial is conducted in Africa, Asia, Europe, Oceania and North America. The aim of this trial is to evaluate the efficacy of activated recombinant human factor VII given in conjunction with standard therapy in the treatment of massive bleeding in subjects with severe blunt and/or penetrating trauma injury.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the subject and/or his/her legally authorised representative (LAR) before any trial-related activities
* Injury(ies) due to a blunt and or penetrating trauma
* Receipt of 6 units of PRBC within a 4 hour period following admittance to the trauma centre
* Receipt of 8 units of PRBC upon administration of trial drug

Exclusion Criteria:

* Prehospital cardiac arrest
* Cardiac arrest in the ER or OR
* Gunshot wound to the head
* Glasgow Coma Scale below 8
* Base deficit of above 15 mEq/l or severe acidosis
* Transfusion of 8 units or more of PRBC prior to arrival in trauma centre

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2002-03; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Number of PRBC (packed red blood cells) units (allogeneic/autologous) transfused

SECONDARY OUTCOMES:
Adverse Events
Changes in coagulation related parameters: APTT (activated partial thromboplastin time), fibrinogen, D-dimers, anti thrombin-III, F1+2 (prothrombin fragment 1+2) and TAT (thrombin anti thrombin complex)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (9):
- Novo Nordisk Investigational Site, Perth, Australia
- Novo Nordisk Investigational Site, Graz, Austria
- Novo Nordisk Investigational Site, Toronto, Ontario, Canada
- Novo Nordisk Investigational Site, Paris, France
- Novo Nordisk Investigational Site, Aachen, Germany
- Novo Nordisk Investigational Site, Jerusalem, Israel
- Novo Nordisk Investigational Site, Singapore, Singapore
- Novo Nordisk Investigational Site, Cape Town, Western Cape, South Africa
- Novo Nordisk Investigational Site, Birmingham, United Kingdom

REFERENCES:
- [Result] Rossaint R, Christensen MC, Choong PI, Boffard KD, Riou B, Rizoli S, Kluger Y, Lefering R, Morris S; NovoSeven(R) Trauma Study Group. Cost-Effectiveness of Recombinant Activated Factor VII as Adjunctive Therapy for Bleeding Control in Severely Injured Trauma Patients in Germany. Eur J Trauma Emerg Surg. 2007 Oct;33(5):528-38. doi: 10.1007/s00068-007-6210-x. Epub 2007 Jul 20. PMID 26814938
- [Result] Boffard KD, Riou B, Warren B, Choong PI, Rizoli S, Rossaint R, Axelsen M, Kluger Y; NovoSeven Trauma Study Group. Recombinant factor VIIa as adjunctive therapy for bleeding control in severely injured trauma patients: two parallel randomized, placebo-controlled, double-blind clinical trials. J Trauma. 2005 Jul;59(1):8-15; discussion 15-8. doi: 10.1097/01.ta.0000171453.37949.b7. PMID 16096533
- [Result] Rizoli SB, Boffard KD, Riou B, Warren B, Iau P, Kluger Y, Rossaint R, Tillinger M; NovoSeven Trauma Study Group. Recombinant activated factor VII as an adjunctive therapy for bleeding control in severe trauma patients with coagulopathy: subgroup analysis from two randomized trials. Crit Care. 2006;10(6):R178. doi: 10.1186/cc5133. PMID 17184516
- [Result] Morris S, Ridley S, Munro V, Christensen MC. Cost effectiveness of recombinant activated factor VII for the control of bleeding in patients with severe blunt trauma injuries in the United Kingdom. Anaesthesia. 2007 Jan;62(1):43-52. doi: 10.1111/j.1365-2044.2006.04896.x. PMID 17156226
- [Result] Champion HR, Fingerhut A, Escobar MA, Weiskopf RB. The role of data and safety monitoring in acute trauma resuscitation research. J Am Coll Surg. 2007 Jan;204(1):73-83. doi: 10.1016/j.jamcollsurg.2006.10.024. PMID 17189115
- [Result] Klitgaard T, Tabanera y Palacios R, Boffard KD, Iau PT, Warren B, Rizoli S, Rossaint R, Kluger Y, Riou B; NovoSeven Trauma Study Group. Pharmacokinetics of recombinant activated factor VII in trauma patients with severe bleeding. Crit Care. 2006;10(4):R104. doi: 10.1186/cc4977. PMID 16859505
- [Result] Kluger Y, Riou B, Rossaint R, Rizoli SB, Boffard KD, Choong PI, Warren B, Tillinger M. Safety of rFVIIa in hemodynamically unstable polytrauma patients with traumatic brain injury: post hoc analysis of 30 patients from a prospective, randomized, placebo-controlled, double-blind clinical trial. Crit Care. 2007;11(4):R85. doi: 10.1186/cc6092. PMID 17686152
- [Result] Hsia CC, Chin-Yee IH, McAlister VC. Use of recombinant activated factor VII in patients without hemophilia: a meta-analysis of randomized control trials. Ann Surg. 2008 Jul;248(1):61-8. doi: 10.1097/SLA.0b013e318176c4ec. PMID 18580208
- [Result] Levy JH, Fingerhut A, Brott T, Langbakke IH, Erhardtsen E, Porte RJ. Recombinant factor VIIa in patients with coagulopathy secondary to anticoagulant therapy, cirrhosis, or severe traumatic injury: review of safety profile. Transfusion. 2006 Jun;46(6):919-33. doi: 10.1111/j.1537-2995.2006.00824.x. PMID 16734808
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com